CLINICAL TRIAL: NCT04238338
Title: Association of Monocyte / Lymphocyte Ratio With Risk of Death and Cardiovascular Events in Peritoneal Dialysis Patients
Brief Title: Association of MLR With Risk of Death and Cardiovascular Events in PD Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Jun Zhang
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2021-08

CONDITIONS: Peritoneal Dialysis; Inflammation
Keywords: monocyte / lymphocyte ratio; peritoneal dialysis; cardiovascular disease; Inflammation; death
MeSH Terms: conditions — Inflammation; Cardiovascular Diseases; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- high MLR group: Divided into high MLR group and low MLR group according to the median of monocyte / lymphocyte ratio(MLR).
  Patients undergo peritoneal dialysis 3, 4 or 5 times per day, with a daily peritoneal dialysate dose of approximately 6000-10000 ml. The glucose concentration of peritoneal dialysate varies depending on the specific requirements of the individual patient for ultrafiltration volume. Three concentrations of glucose peritoneal dialysis solution are available for peritoneal dialysis patients. The low concentration is 1.5% or 2.5% and the high concentration is 4.25%. In principle, a 1.5% glucose peritoneal dialysis solution is first applied, or a high concentration of 4.25% glucose peritoneal dialysis solution can be appropriately applied according to the actual situation. Other drugs continued to be used in patients with other diseases.
  Interventions: Other: monocyte / lymphocyte ratio
- low MLR group: Divided into high MLR group and low MLR group according to the median of monocyte / lymphocyte ratio(MLR).
  Patients undergo peritoneal dialysis 3, 4 or 5 times per day, with a daily peritoneal dialysate dose of approximately 6000-10000 ml. The glucose concentration of peritoneal dialysate varies depending on the specific requirements of the individual patient for ultrafiltration volume. Three concentrations of glucose peritoneal dialysis solution are available for peritoneal dialysis patients. The low concentration is 1.5% or 2.5% and the high concentration is 4.25%. In principle, a 1.5% glucose peritoneal dialysis solution is first applied, or a high concentration of 4.25% glucose peritoneal dialysis solution can be appropriately applied according to the actual situation. Other drugs continued to be used in patients with other diseases.
  Interventions: Other: monocyte / lymphocyte ratio

INTERVENTIONS:
Other: monocyte / lymphocyte ratio — The lymphocyte / monocyte ratio should be tested every 3-6months after the start of the study, and the final value is the average

SUMMARY:
The current incidence of chronic kidney disease (CKD) in China is approximately 10.8%, with approximately 119 million patients. Among them, patients with end-stage renal disease (ESRD) are about 200-250 cases per million population. At present, the main renal replacement therapy is: hemodialysis (HD) or peritoneal dialysis (PD). Compared with HD, PD is easy to operate, better preserves residual renal function, has early survival advantages, and is more cost-effective. Despite this, the prognosis of PD patients is still not ideal, and cardiovascular disease (CVD) remains the leading cause of death in PD patients. Persistent inflammatory states are critical in the pathogenesis of CVD such as atherosclerosis and vascular calcification, and lead to protein energy expenditure and premature death outcomes in patients with CKD. Therefore, screening for markers that predict the risk of CVD in dialysis patients is essential. Some novel inflammatory markers have been shown to have diagnostic and prognostic value in ESRD patients in terms of inflammation, malnutrition, cardiovascular calcification, all-cause, and risk of CVD death. Among them, blood cell related parameters such as neutrophil / lymphocyte ratio (NLR) and monocyte / lymphocyte ratio (MLR)can reflect both inflammation and immune deficiency. NLR, MLR has been proposed as a new inflammatory biomarker and a potential predictor of cardiovascular risk. Studies have reported that MLR is associated with cardiovascular death and all-cause death risk in hemodialysis patients, and is superior to NLR. However, the relationship between MLR and the prognosis of patients with peritoneal dialysis is rarely reported. Therefore, in this study, we aimed to evaluate the association of MLR with risk of death and cardiovascular events in PD patients.

DETAILED DESCRIPTION:
The epidemiological survey of chronic kidney disease in China shows that the current incidence of chronic kidney disease (CKD) in China is about 10.8%, with about 119 million patients. About 2% of patients will enter the stage of end-stage renal disease (ESRD) and require dialysis or kidney transplantation to support life. Currently the main renal replacement therapy is: hemodialysis (HD) or peritoneal dialysis (PD). Among them, PD patients are increasing year by year. As of 2016, more than 900,000 people in Asia are undergoing maintenance dialysis (218 cases per million population). Statistics from the CNRDS system show that as of the end of 2017, the number of PD patients in China has reached 86264. Compared with HD, PD is easy to operate, better preserves residual renal function, has early survival advantages, and is more cost-effective. In spite of this, the prognosis of PD patients is still unsatisfactory. At present, the main causes of death in PD patients are cardiovascular disease, peritoneal dialysis-related peritonitis, gastrointestinal bleeding, and tumors. Among them, cardiovascular disease (CVD) is the most important, accounting for about 50% of the deaths of PD patients. Among all CVD events, coronary heart disease, heart failure, and stroke are the most common. CVD risk factors for dialysis patients can be divided into traditional and non-traditional categories. Traditional Framingham risk factors can only explain some of the CVD risks of PD patients. Non-traditional risk factors, especially persistent inflammatory states, are essential in the pathogenesis of CVD such as atherosclerosis and vascular calcification, and lead to protein energy expenditure and premature death outcomes in patients with CKD.

The causes of chronic inflammation in patients with peritoneal dialysis are mainly divided into two aspects. Dialysis-related factors include: catheter-related infections, continuous exposure to biologically incompatible PD solutions, peritonitis, increased adipose tissue, and adipose factor balance disorders; associated with low GFR Factors include decreased clearance of pro-inflammatory factors, accumulation of uremic toxins, endotoxin exposure, oxidative stress, increased volume load, oral or other organ infections, and susceptibility to infections. The causes of inflammation in peritoneal dialysis are interconnected, leading to a persistent state of inflammation that ultimately increases the risk of cardiovascular events. Therefore, it is important to screen for markers that predict the risk of CVD in dialysis patients. At present, various inflammatory mediators, such as c-reactive protein（CRP）, interleukins（IL）and tumor necrosis factor（TNF）, have been studied and proven to independently predict the risk of CVD in dialysis patients. CRP can induce the expression of adhesion molecules in endothelial cells, increase the adhesion of vascular endothelial cells and monocytes; promote the formation of foam cells and atherosclerosis; aggravate vascular endothelial dysfunction; TNF-α can increase the expression and activity of alkaline phosphatase, enhance Isolated vascular wall calcification; aggravates vascular endothelial dysfunction; promotes left ventricular remodeling and aggravates left ventricular dysfunction. IL-6 can stimulate macrophages to secrete monocyte chemotactic protein 1, induce endothelial cell adhesion molecule expression; stimulate vascular smooth muscle cell proliferation and migration; aggravate vascular endothelial dysfunction; and induce cardiac hypertrophy. Although the mechanisms are different, they all increase the risk of CVD death in dialysis patients by aggravating vascular endothelial dysfunction, promoting ventricular remodeling and inducing myocardial hypertrophy. However, such markers are expensive and their detection is not easy to limit their clinical application. This prompted researchers to devote themselves to mining new markers of inflammation. In recent years, experts and scholars have become interested in blood cell parameters. Previous studies have shown that white blood cells and their subgroups (neutrophils, lymphocytes, monocytes) ), Neutrophil / lymphocyte ratio (NLR), monocyte / lymphocyte ratio (MLR), platelet / lymphocyte ratio (PLR) and other indicators have important predictive value for all causes and prognosis of cardiovascular disease in dialysis population . They have the advantages of low cost and easy detection. Among them, MLR has been proven to be an independent predictor of death in cardiovascular diseases such as coronary heart disease and heart failure. Previous research found. Monocytes play a key role in the occurrence and development of atherosclerosis. After the initial injury, endothelial cells are activated and promote monocytes to roll, attach and migrate under the endothelium. Monocytes that migrate to the subendothelium can differentiate into dendritic cells, which are key participants in activating adaptive immunity, or differentiate into macrophages, which secrete pro-inflammatory cytokines, thereby recruiting more immune cells and Promote inflammation. Macrophage phagocytosis of lipoprotein particles can lead to the formation of fatty streaks, the earliest ultrastructural changes in the formation of atherosclerosis. The migration of smooth muscle cells from the medial membrane to the intimal membrane further promotes the atherogenic process. Monocyte-derived cells transform this early lesion into advanced atherosclerotic plaques, which contain lipid-rich and macrophage-rich necrotic cores that eventually cause the plaque to rupture. In addition, previous studies have shown that physiological stress can lead to a significant increase in systemic cortisol production, which has led to a shift in leukocyte differentiation toward a decrease in lymphocytes and an increase in the percentage of granulocytes. Measuring lymphocyte counts can reflect stress levels. In patients with coronary heart disease, studies have shown that a decrease in lymphocyte count is an independent predictor of prognosis in patients with coronary heart disease; there is a phenomenon of lymphocyte apoptosis on the endothelium of atherosclerotic injured blood vessels. Therefore, low lymphocytes can reflect the occurrence and development of atherosclerotic diseases. In patients with end-stage renal disease, there will be changes in the number of immune cells such as increased monocytes and decreased lymphocytes. First, the decline in renal function causes retention of uremic toxins and cytokines, which leads to increased proinflammatory cytokines and oxidative stress. It further stimulates the proliferation of monocytes, and at the same time down-regulates immunity, resulting in a decrease in the number and function of lymphocytes, which in turn promotes inflammation and oxidative stress, and continues a vicious cycle. MLR can integrate pro-inflammatory and anti-inflammatory effects, and simultaneously reflect inflammation and immune deficiency. It may be an important marker of inflammation in patients with end-stage renal disease. In 2017, Xiang F et al. For the first time found in a prospective cohort study of 355 hemodialysis patients that high MLR levels were independent predictors of all-cause and CVD mortality in hemodialysis patients, and exceeded the predictive value of NLR However, there are no reports about MLR and prognosis in patients with peritoneal dialysis at home and abroad. Our previous retrospective analysis showed that the all-cause and cardiovascular disease survival rates of patients in the low MLR group were significantly higher than those in the high MLR group; high MLR levels were associated with all-cause and increased risk of cardiovascular death in patients with peritoneal dialysis. However, because retrospective studies cannot determine causality, there may be problems such as selection bias. Therefore, a prospective, large-sample study is needed to further explore the correlation between MLR and the prognosis of PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent continuous ambulatory peritoneal dialysis for at least 3 months.

Exclusion Criteria:

* Age <18 years, with acute or chronic infections such as lung infection,peritoneal dialysis-related peritonitis, urinary system infection, etc .
* With history of malignant tumor or blood disease.
* With rheumatic immune diseases, such as systemic lupus erythematosus, vasculitis , Sjögren's syndrome, etc .
* Used immunosuppressants, such as glucocorticoids, calcineurin inhibitors, etc .
* Women during pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent continuous ambulatory peritoneal dialysis in the Department of Nephrology of Southern Medical University Zhujiang Hospital，and voluntarily signed informed consent to join the study.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality and cardiovascular mortality | 12 months
  Proportion of all-cause and cardiovascular deaths during follow-up

SECONDARY OUTCOMES:
The Incidence of cardiovascular events | 12 months
  Cardiovascular events during follow-up (including acute heart failure, angina, acute myocardial infarction, arrhythmias requiring treatment, transient ischemic attack (TIA), cerebral infarction or cerebral hemorrhage, peripheral vascular disease)
The Incidence of peritoneal dialysis-associated peritonitis | 12 months
  Peritoneal dialysis-related peritonitis refers to the complications of peritonitis such as abdominal pain, fever, or turbid dialysate during peritoneal dialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Doctor, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) is not available.

REFERENCES:
- [Background] Lameire N, Van Biesen W. Epidemiology of peritoneal dialysis: a story of believers and nonbelievers. Nat Rev Nephrol. 2010 Feb;6(2):75-82. doi: 10.1038/nrneph.2009.210. Epub 2009 Dec 15. PMID 20010897
- [Background] Li PK, Chow KM, Van de Luijtgaarden MW, Johnson DW, Jager KJ, Mehrotra R, Naicker S, Pecoits-Filho R, Yu XQ, Lameire N. Changes in the worldwide epidemiology of peritoneal dialysis. Nat Rev Nephrol. 2017 Feb;13(2):90-103. doi: 10.1038/nrneph.2016.181. Epub 2016 Dec 28. PMID 28029154
- [Background] Saran R, Steffick D, Bragg-Gresham J. The China Kidney Disease Network (CK-NET): "Big Data-Big Dreams". Am J Kidney Dis. 2017 Jun;69(6):713-716. doi: 10.1053/j.ajkd.2017.04.008. No abstract available. PMID 28532632
- [Background] Cho Y, Hawley CM, Johnson DW. Clinical causes of inflammation in peritoneal dialysis patients. Int J Nephrol. 2014;2014:909373. doi: 10.1155/2014/909373. Epub 2014 May 6. PMID 24895536
- [Background] Akchurin OM, Kaskel F. Update on inflammation in chronic kidney disease. Blood Purif. 2015;39(1-3):84-92. doi: 10.1159/000368940. Epub 2015 Jan 20. PMID 25662331
- [Background] Miyamoto T, Carrero JJ, Stenvinkel P. Inflammation as a risk factor and target for therapy in chronic kidney disease. Curr Opin Nephrol Hypertens. 2011 Nov;20(6):662-8. doi: 10.1097/MNH.0b013e32834ad504. PMID 21825982
- [Background] Li PK, Ng JK, Mcintyre CW. Inflammation and Peritoneal Dialysis. Semin Nephrol. 2017 Jan;37(1):54-65. doi: 10.1016/j.semnephrol.2016.10.007. PMID 28153195
- [Background] Carrero JJ, Stenvinkel P. Inflammation in end-stage renal disease--what have we learned in 10 years? Semin Dial. 2010 Sep-Oct;23(5):498-509. doi: 10.1111/j.1525-139X.2010.00784.x. PMID 21039875
- [Background] Miller LM, Sood MM, Sood AR, Reslerova M, Komenda P, Rigatto C, Bueti J. Cardiovascular disease in end-stage renal disease: the challenge of assessing and managing cardiac disease in dialysis patients. Int Urol Nephrol. 2010 Dec;42(4):1007-14. doi: 10.1007/s11255-010-9857-x. Epub 2010 Oct 20. PMID 20960231
- [Background] Jegatheesan D, Cho Y, Johnson DW. Clinical Studies of Interventions to Mitigate Cardiovascular Risk in Peritoneal Dialysis Patients. Semin Nephrol. 2018 May;38(3):277-290. doi: 10.1016/j.semnephrol.2018.02.007. PMID 29753403
- [Background] Wang AY, Brimble KS, Brunier G, Holt SG, Jha V, Johnson DW, Kang SW, Kooman JP, Lambie M, McIntyre C, Mehrotra R, Pecoits-Filho R. ISPD Cardiovascular and Metabolic Guidelines in Adult Peritoneal Dialysis Patients Part I - Assessment and Management of Various Cardiovascular Risk Factors. Perit Dial Int. 2015 Jul-Aug;35(4):379-87. doi: 10.3747/pdi.2014.00279. PMID 26228782
- [Background] Liakopoulos V, Roumeliotis S, Gorny X, Eleftheriadis T, Mertens PR. Oxidative Stress in Patients Undergoing Peritoneal Dialysis: A Current Review of the Literature. Oxid Med Cell Longev. 2017 Dec 27;2017:3494867. doi: 10.1155/2017/3494867. eCollection 2017. PMID 29750088
- [Background] Saxena AB. Recent advances in the management of peritoneal dialysis patients. F1000Prime Rep. 2015 May 1;7:57. doi: 10.12703/P7-57. eCollection 2015. PMID 26097730
- [Background] Betjes MG. Immune cell dysfunction and inflammation in end-stage renal disease. Nat Rev Nephrol. 2013 May;9(5):255-65. doi: 10.1038/nrneph.2013.44. Epub 2013 Mar 19. PMID 23507826
- [Background] Ernandez T, Mayadas TN. The Changing Landscape of Renal Inflammation. Trends Mol Med. 2016 Feb;22(2):151-163. doi: 10.1016/j.molmed.2015.12.002. Epub 2016 Jan 7. PMID 26778189
- [Background] Johnson DW, Wiggins KJ, Armstrong KA, Campbell SB, Isbel NM, Hawley CM. Elevated white cell count at commencement of peritoneal dialysis predicts overall and cardiac mortality. Kidney Int. 2005 Feb;67(2):738-43. doi: 10.1111/j.1523-1755.2005.67135.x. PMID 15673324
- [Background] Li H, Lu X, Xiong R, Wang S. High Neutrophil-to-Lymphocyte Ratio Predicts Cardiovascular Mortality in Chronic Hemodialysis Patients. Mediators Inflamm. 2017;2017:9327136. doi: 10.1155/2017/9327136. Epub 2017 Feb 21. PMID 28316378
- [Background] Xiang F, Chen R, Cao X, Shen B, Liu Z, Tan X, Ding X, Zou J. Monocyte/lymphocyte ratio as a better predictor of cardiovascular and all-cause mortality in hemodialysis patients: A prospective cohort study. Hemodial Int. 2018 Jan;22(1):82-92. doi: 10.1111/hdi.12549. Epub 2017 Apr 12. PMID 28403540
- [Background] Hou H, Sun T, Li C, Li Y, Guo Z, Wang W, Li D. An overall and dose-response meta-analysis of red blood cell distribution width and CVD outcomes. Sci Rep. 2017 Feb 24;7:43420. doi: 10.1038/srep43420. PMID 28233844
- [Background] Saionji K, Ohsaka A. Expansion of CD4+CD16+ blood monocytes in patients with chronic renal failure undergoing dialysis: possible involvement of macrophage colony-stimulating factor. Acta Haematol. 2001;105(1):21-6. doi: 10.1159/000046528. PMID 11340249
- [Background] Laudanski K, Nowak Z. Aberrant function and differentiation of monocytes in end stage renal disease. Arch Immunol Ther Exp (Warsz). 2012 Dec;60(6):453-9. doi: 10.1007/s00005-012-0191-0. Epub 2012 Oct 19. PMID 23080050
- [Background] Turkmen K, Guney I, Yerlikaya FH, Tonbul HZ. The relationship between neutrophil-to-lymphocyte ratio and inflammation in end-stage renal disease patients. Ren Fail. 2012;34(2):155-9. doi: 10.3109/0886022X.2011.641514. Epub 2011 Dec 16. PMID 22172001
- [Background] Afari ME, Bhat T. Neutrophil to lymphocyte ratio (NLR) and cardiovascular diseases: an update. Expert Rev Cardiovasc Ther. 2016;14(5):573-7. doi: 10.1586/14779072.2016.1154788. Epub 2016 Mar 4. PMID 26878164
- [Background] Agarwal R, Light RP. Patterns and prognostic value of total and differential leukocyte count in chronic kidney disease. Clin J Am Soc Nephrol. 2011 Jun;6(6):1393-9. doi: 10.2215/CJN.10521110. Epub 2011 May 5. PMID 21551023
- [Background] Kim JH, Lim S, Park KS, Jang HC, Choi SH. Total and differential WBC counts are related with coronary artery atherosclerosis and increase the risk for cardiovascular disease in Koreans. PLoS One. 2017 Jul 28;12(7):e0180332. doi: 10.1371/journal.pone.0180332. eCollection 2017. PMID 28753607
- [Background] Heine GH, Ortiz A, Massy ZA, Lindholm B, Wiecek A, Martinez-Castelao A, Covic A, Goldsmith D, Suleymanlar G, London GM, Parati G, Sicari R, Zoccali C, Fliser D; European Renal and Cardiovascular Medicine (EURECA-m) working group of the European Renal Association-European Dialysis and Transplant Association (ERA-EDTA). Monocyte subpopulations and cardiovascular risk in chronic kidney disease. Nat Rev Nephrol. 2012 Mar 13;8(6):362-9. doi: 10.1038/nrneph.2012.41. PMID 22410492
- [Background] Kanbay M, Solak Y, Unal HU, Kurt YG, Gok M, Cetinkaya H, Karaman M, Oguz Y, Eyileten T, Vural A, Covic A, Goldsmith D, Turak O, Yilmaz MI. Monocyte count/HDL cholesterol ratio and cardiovascular events in patients with chronic kidney disease. Int Urol Nephrol. 2014 Aug;46(8):1619-25. doi: 10.1007/s11255-014-0730-1. Epub 2014 May 23. PMID 24853998
- [Background] Pereira R, Costa E, Goncalves M, Miranda V, do Sameiro Faria M, Quintanilha A, Belo L, Lima M, Santos-Silva A. Neutrophil and monocyte activation in chronic kidney disease patients under hemodialysis and its relationship with resistance to recombinant human erythropoietin and to the hemodialysis procedure. Hemodial Int. 2010 Jul;14(3):295-301. doi: 10.1111/j.1542-4758.2010.00450.x. PMID 20649681
- [Background] Turkmen K, Erdur FM, Ozcicek F, Ozcicek A, Akbas EM, Ozbicer A, Demirtas L, Turk S, Tonbul HZ. Platelet-to-lymphocyte ratio better predicts inflammation than neutrophil-to-lymphocyte ratio in end-stage renal disease patients. Hemodial Int. 2013 Jul;17(3):391-6. doi: 10.1111/hdi.12040. Epub 2013 Mar 24. PMID 23522328
- [Background] Taymez DG, Ucar E, Turkmen K, Ucar R, Afsar B, Gaipov A, Turk S. The Predictive Value of Platelet/Lymphocyte Ratio in Hemodialysis Patients With Erythropoietin Resistance. Ther Apher Dial. 2016 Apr;20(2):118-21. doi: 10.1111/1744-9987.12380. Epub 2016 Mar 1. PMID 26929254
- [Background] Ommen SR, Gibbons RJ, Hodge DO, Thomson SP. Usefulness of the lymphocyte concentration as a prognostic marker in coronary artery disease. Am J Cardiol. 1997 Mar 15;79(6):812-4. doi: 10.1016/s0002-9149(96)00878-8. PMID 9070569
- [Background] Zouridakis EG, Garcia-Moll X, Kaski JC. Usefulness of the blood lymphocyte count in predicting recurrent instability and death in patients with unstable angina pectoris. Am J Cardiol. 2000 Aug 15;86(4):449-51. doi: 10.1016/s0002-9149(00)00963-2. No abstract available. PMID 10946041